CLINICAL TRIAL: NCT00750763
Title: A Prospective Audit of Tolerability, Mucosal Cleansing Efficacy and Mucosal Abnormalities Associated With Standard Orally Administered Colon Cleansing Preparations for Colonoscopy
Brief Title: Tolerability, Efficacy and Mucosal Inflammation Associated With Orally Administered Colon Cleansing for Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fremantle Hospital and Health Service (Other)
Responsible Party: A/Prof Ian C Lawrance, Department of Gastroenterology, Fremantle Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FHHS
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Colonoscopy
Keywords: Mucosal inflammation; Fleet; Picoprep; Colonlytely; Colonoscopy; tolerability; efficacy
MeSH Terms: conditions — Mucositis | interventions — Polyethylene Glycols; picosulfate sodium; sodium phosphate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): PEG (Colonlytely) - 4 litres
  Interventions: Drug: Colonlytely
- 2 (Active Comparator): Picosulphate (Picolax/Picoprep) - 2 sachets
  Interventions: Drug: Picolax/Picoprep
- 3 (Active Comparator): Sodium Phosphate (Fleet) - 2 bottles
  Interventions: Drug: Fleet

INTERVENTIONS:
Drug: Colonlytely — Bowel preparation
  Other Names: Polyethylene glycol
  Arms: 1
Drug: Picolax/Picoprep — Bowel preparation
  Other Names: Picosulphate
  Arms: 2
Drug: Fleet — Bowel preparation
  Other Names: Sodium Phosphate
  Arms: 3

SUMMARY:
Colonoscopy is the gold standard investigation for assessing the lining of the colon. Colon cleansing preparations are required to be taken prior to colonoscopy to provide effective visualisation and identification of any abnormalities and different types of colon cleansing preparations exist.

Some colon cleansing preparations have been shown to cause visible changes in the lining of the bowel which may cause confusion and incorrect diagnoses to be made.

This audit aims to assess the ability of different colon cleansing preparations to clear the colon of faeces. The tolerability of each will also be assessed, as will any changes in the lining of the bowel to assess if one type of colon preparation is more likely to cause visible changes than another.

DETAILED DESCRIPTION:
There are several published trials of different colon cleansing agents for colonoscopy (which is the investigation of choice for visualisation of the colonic mucosa) which compare different regimens. However, a recent published meta-analysis has shown that most audits and studies were underpowered with poor study design and so no consensus on the most effective preparation exists1. 10-20% of failed colonoscopy is attributable to inadequate bowel cleansing which has a negative impact on the detection of potential malignant lesions in the colon3 as well as requiring the patient to attend again for further colonoscopy after repeated colon cleansing which also impacts on waiting lists and healthcare costs.

Colon cleansing preparations can be broadly classified into three groups. Osmotic laxatives such as sodium phosphate (NaP) increase colon water content by attracting extracellular fluid efflux through the bowel wall. Polyethylene glycol (PEG) laxatives are high molecular weight non-absorbable polymers that are administered in a dilute electrolyte solution, this is retained in the colon where it acts as a bowel cleanser without any significant fluid exchange across the colonic mucosa. The third group are stimulant laxatives such as senna or sodium picosulphate which work primarily by enhancing smooth muscle contractility and also they may increase bowel water content.

Previous published audits and studies comparing different types of colon cleansing preparations have been limited by small sample size with only 5 published papers having over 100 patients in each arm of the study. These 5 studies suggest that NaP may be better than PEG but the recent meta-analysis failed to show this, primarily due to the large number of smaller studies showing PEG was better than NaP. Interpretation of the studies is limited by inconsistent and poorly defined measures of efficacy outcome. Most studies have used a subjective endoscopists assessment of the overall quality of the bowel preparation making comparisons between studies impossible. Recently a calibrated externally validated outcome assessment tool has been developed to objectively quantify the quality of bowel preparation4, but no randomised published study has yet utilised this tool.

In the absence of clear difference in efficacy between preparations then patient tolerability is likely to be an important distinguishing feature when selecting a treatment. Data on tolerability outcomes is limited but there is some evidence that PEG solutions are less well tolerated due to the volume of liquid required to drink. This is an area where further study is needed.

The ability of a colonic cleansing preparation to clean the colon effectively also must be balanced by its ability to not induce changes in the lining of the bowel itself. Ulceration and inflammation of the colon has been shown to occur in 3-24% of patients using NaP compared with 1-2% in those receiving PEG. Such findings can be mistaken for inflammatory bowel disease such as Crohns or put down to drug induced changes such as non steroidal anti inflammatory agents (NSAIDs). However, these studies have been either non randomised5 or underpowered to detect real differences.

The most satisfactory colonic cleansing agent in terms of efficacy, tolerability and safety therefore remains unclear.

The aims of the project are:

1. To assess which bowel preparation provides the best colon cleansing using a validated score.
2. To assess the incidence of mucosal inflammation/ulceration induced by each colon cleansing agent.
3. To see which colon cleansing agent is best tolerated by patients.

The information gained from this audit will enable the type of colonic cleansing preparation to be tailored to the subjects indication for requiring colonoscopy. For example in those with possible inflammatory bowel disease the colon cleansing agent which produces the least mucosal inflammation would be required to reduce the incidence of a false positive diagnosis whilst the colon cleansing agent which is most tolerable may be more important in the elderly.

This study will be a prospective blinded audit comparing three colon cleansing agents, which are used routinely in clinical practice for colonoscopy. The three will be Sodium Phosphate (Fleet), Sodium Picosulphate (Picolax/Picoprep) and PEG (Colonlytlye).

All patients who are referred to undergo colonoscopy would be entered into the study except for:

1. Prior history of inflammatory bowel disease or suspected inflammatory bowel disease, or patients on current non steroidal antiinflammatory medication (excluding low dose aspirin). These patients may have mucosal inflammation/ulceration which would prevent analysis of mucosal abnormalities due to the colon cleansing agent and so would not be studied.
2. Patients with heart failure (NYHA >2) or renal failure (GFR<30) (since fluid shifts associated with sodium phosphate bowel preparation have been reported).
3. All patients over the age of 75 due to potential dehydration and hyperphosphatemia from the bowel preparations.

Each patient would be randomised to receive one of the three colon cleansing agents (Sodium Phosphate, Sodium Picosulphate or PEG) that are routinely used in clinical practice. The endoscopy administration staff at each site would be responsible for random allocation of the bowel preparation using random number generation with the resultant bowel preparation being collected by the patient from a pharmacy, as per usual practice, prior to the colonoscopy. There are no exclusion criteria for bowel preparation selection.

On the day of colonoscopy but prior to the procedure an assessment of the tolerability of the colon cleansing agent would be made using a questionnaire.

During colonoscopy an assessment of the efficacy of the colon cleansing agent is made by the blinded colonoscopist using the previously validated Ottawa bowel preparation assessment tool.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are referred to undergo ambulatory colonoscopy at Kaleeya Hospital would be entered into the study

Exclusion Criteria:

* Prior history of inflammatory bowel disease or suspected inflammatory bowel disease, or patients on current non steroidal antiinflammatory medication (excluding low dose aspirin). These patients may have mucosal inflammation/ulceration which would prevent analysis of mucosal abnormalities due to the colon cleansing agent and so would not be studied.
* Patients with heart failure (NYHA >2) or renal failure (GFR<30) (since fluid shifts associated with sodium phosphate bowel preparation have been reported).
* All patients over the age of 75 due to potential dehydration and hyperphosphatemia from the bowel preparations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To assess which bowel preparation provides the best colon cleansing using a validated score and is best tolerated by patients. | At time of colonoscopy

SECONDARY OUTCOMES:
To assess the incidence of mucosal inflammation/ulceration induced by each colon cleansing agent. | At time of colonscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ian C Lawrance, MD PhD, Principal Investigator — Department of Gastroenterology, Fremantle Hospital
Locations (1):
- Department of Gastroenterology, Fremantle Hospital, Fremantle, Western Australia, Australia

REFERENCES:
- [Derived] Lawrance IC, Willert RP, Murray K. A validated bowel-preparation tolerability questionnaire and assessment of three commonly used bowel-cleansing agents. Dig Dis Sci. 2013 Apr;58(4):926-35. doi: 10.1007/s10620-012-2449-0. Epub 2012 Oct 25. PMID 23095990
- [Derived] Lawrance IC, Willert RP, Murray K. Bowel cleansing for colonoscopy: prospective randomized assessment of efficacy and of induced mucosal abnormality with three preparation agents. Endoscopy. 2011 May;43(5):412-8. doi: 10.1055/s-0030-1256193. Epub 2011 May 4. PMID 21547879